CLINICAL TRIAL: NCT00385177
Title: A Multicenter Phase 1 Dose Escalation Study of SN2310 Injectable Emulsion in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Dose Escalation Study of SN2310 Injectable Emulsion in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-2310-06-101
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Pelvic Neoplasms; Lung Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Pelvic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): SN2310 Injectable Emulsion
  Interventions: Drug: SN2310 Injectable Emulsion

INTERVENTIONS:
Drug: SN2310 Injectable Emulsion — Escalating doses given IV every three weeks

SUMMARY:
This is a Phase 1 open-label study of SN2310 Injectable Emulsion in patients with advanced solid malignancies. The study is designed to determine the maximum tolerated dose and dose-limiting toxicity of SN2310 Injectable Emulsion, and to characterize the pharmacokinetics of SN2310 and SN-38 following intravenous administration of SN2310 Injectable Emulsion. Additionally, evaluation of side effects as a function of dose, and observation of any anti-tumor effects of SN2310 Injectable Emulsion will be made.

DETAILED DESCRIPTION:
This is a Phase 1 open-label study of SN2310 Injectable Emulsion in patients with advanced solid malignancies who have failed conventional therapy. SN2310 Injectable Emulsion will be administered intravenously every 21 days. The study is designed to determine the maximum tolerated dose and dose-limiting toxicity of SN2310 Injectable Emulsion; to characterize the pharmacokinetics of SN2310 and SN-38 following intravenous administration of SN2310 Injectable Emulsion; to evaluate side effects as a function of dose level; and, to observe any anti-tumor effects of SN2310 Injectable Emulsion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of solid tumor with disease progression despite standard therapy and/or for which no other solid therapeutic option exists
* ANC > 1,500 cell/mm3, platelets > 100,000/mm3 and Hgb > 9 g/dl
* At least one unidimensionally measurable lesion per RECIST
* Negative serum or urine pregnancy test, if female of childbearing potential

Exclusion Criteria:

* Female who is pregnant or lactating
* History of chronic diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | December 2008
Dose-Limiting Toxicity | December 2008
Adverse Events | December 2008
Pharmacokinetic parameters for SN2310 and SN-38 | December 2008

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee